CLINICAL TRIAL: NCT05664061
Title: A Phase III, Randomized, Multicenter, Parallel-group Clinical Trial for Examining the Therapeutic Equivalence Between Fluticasone Propionate 100 mcg and Salmeterol 50 mcg Inhalation Powder/Respirent Pharmaceuticals vs. ADVAIR DISKUS® 100/50 mcg Inhalation Powder/GSK in Patients With Asthma
Brief Title: Bioequivalence With Clinical Endpoint Study of Fluticasone Propionate 100 mcg and Salmeterol 50 mcg Inhalation Powder/Respirent Pharmaceuticals vs. ADVAIR DISKUS® 100/50 mcg Inhalation Powder/GSK in Patients With Asthma
Acronym: AERO-PD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Respirent Pharmaceuticals Co Ltd. (Industry)
Collaborators: Becro Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BECRO/RESP/AERO-PD
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Asthma
Keywords: asthma; therapeutic equivalence; bioequivalence; fluticasone propionate; salmeterol
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: observer-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Fluticasone propionate 100 mcg and Salmeterol 50 mcg inhalation powder/Respirent Pharmaceuticals (Experimental): Test (T)
  Interventions: Drug: Fluticasone Propionate 100 mcg and Salmeterol 50 mcg inhalation Powder/Respirent Pharmaceuticals
- ADVAIR DISKUS® 100/50 mcg inhalation powder pre-dispensed/GSK (Active Comparator): Reference (R)
  Interventions: Drug: ADVAIR DISKUS® 100/50 mcg inhalation powder pre-dispensed/GSK
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone Propionate 100 mcg and Salmeterol 50 mcg inhalation Powder/Respirent Pharmaceuticals — twice daily inhalation throughout the treatment period
  Other Names: Test (T)
  Arms: Fluticasone propionate 100 mcg and Salmeterol 50 mcg inhalation powder/Respirent Pharmaceuticals
Drug: ADVAIR DISKUS® 100/50 mcg inhalation powder pre-dispensed/GSK — twice daily inhalation throughout the treatment period
  Other Names: Refernce (R)
  Arms: ADVAIR DISKUS® 100/50 mcg inhalation powder pre-dispensed/GSK
Drug: Placebo — twice daily inhalation throughout the treatment period
  Arms: Placebo

SUMMARY:
Τherapeutic equivalence, randomized, multiple-dose, placebo-controlled, observer-blind, parallel group design consisting of a 2-week run-in period followed by a 4-week treatment period with Fluticasone propionate 100 mcg and Salmeterol 50 mcg inhalation powder/Respirent Pharmaceuticals (Test) or ADVAIR DISKUS® 100/50 mcg (Reference) or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects (≥12 years of age) of non-childbearing or of childbearing potential committed to consistent and correct use of an acceptable method of birth control.
2. Patients diagnosed with asthma, as defined by the National Asthma Education and Prevention Program (NAEPP), at least 12 weeks prior to screening.
3. Pre-bronchodilator FEV1 of ≥40% and ≤85% of the predicted value (for age ≥18 years), or ≥65% and ≤90% predicted normal value (for ages 12 to 17 years) during the screening visit and on the first day of treatment.
4. Currently non-smoking; had not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and had ≤ 10 pack-years of historical use.
5. ≥12% and 200 mL reversibility of FEV1 within 30 minutes following 400 mcg salbutamol (4 puffs) inhalation (pMDI). This may be demonstrated at the Screening Visit or this test may be repeated on a different day if the patient fails the first attempt anytime in the period leading up to Visit 2 (randomization); If reversibility is not demonstrated up to Visit 2 then patients may be permitted to enter the study with historical evidence of reversibility that was performed within 2 years prior to Visit 1 and patients should be stable on their chronic asthma treatment regimen for at least 4 weeks prior to enrolment.
6. Patients who are able to discontinue their asthma medications (inhaled corticosteroids and long-acting β agonists) during the run-in period and for remainder of the study, according to investigator's judgement.
7. Patients who are able to replace current short-acting β agonists (SABAs) with salbutamol inhaler for use as needed for the duration of the study (subjects should be able to withhold all inhaled SABAs for at least 6 hours prior to lung function assessments on study visits).
8. Patients who are able to continue treatment with theophylline or montelukast without a significant adjustment of dosage, formulation, dosing interval for the duration of the study, and judged able by the investigator to withhold them for the specified minimum time intervals prior to each patient visit: 1) montelukast 36 hours 2) short-acting forms of theophylline 12 hours, 3) twice-a-day controlled-release forms of theophylline 24 hours, 4) once-a-day controlled-release forms of theophylline 36 hours.
9. Patients who are able to understand the requirements of the clinical trial and to agree to return for the required follow-up visits.
10. Willing to provide voluntary written informed consent and data protection declaration (and in the case of a minor their parent/guardian was able to give) before any clinical trial related procedure is performed.

Exclusion Criteria:

1. Life-threatening asthma, defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnia; respiratory arrest or hypoxic seizures, asthma related syncopal episode(s), or hospitalizations within the past year to the screening or during the run-in period.
2. Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia.
3. Historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbated during the study.
4. Hypersensitivity to any sympathomimetic drug (e.g., salmeterol/albuterol) or to any inhaled, intranasal, or systemic corticosteroid therapy.
5. History of hypersensitivity to lactose
6. Medication(s) with the potential to affect the course of asthma or to interact with sympathomimetic amines, e.g.: β-blockers, oral decongestants, benzodiazepines, digitalis, phenothiazines, polycyclic antidepressants, monoamine oxidase inhibitors.
7. symptoms or signs of viral or bacterial, upper or lower respiratory tract infection or sinus or middle ear infection within 4 weeks prior to the screening visit or during the run-in period.
8. Asthma exacerbation (i.e. acute or sub-acute worsening in symptoms and lung function from the patient's usual status) within 6 weeks prior to the screening visit or during the run-in period
9. Use of oral or parenteral corticosteroids within 4 weeks prior to Screening visit (Visit 1)
10. Factors (e.g., infirmity, disability or geographic location) that the investigator felt would likely limit the patient's compliance with the study protocol or scheduled clinic visits.
11. Female Subjects who are pregnant or breastfeeding.
12. Women of child-bearing age that are not surgically incapable of pregnancy and are not willing to use an acceptable method of birth control.
13. Current participation or not yet completed period of at least 30 days since ending other investigational device or drug trial(s).
14. Unwillingness or inability to comply with the clinical trial procedures;
15. Unwillingness to consent to storage, saving and transmission of pseudonymous medical data for clinical trial reasons;
16. Who are legally incapacitated;
17. Who are legally detained in an official institute.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
FEV1 AUC (0-12h) | 12 hours
  Area under the serial FEV1(L)-time curve calculated from time zero to 12 hours (AUC0-12h) on the first day of the treatment after adjustment for baseline (change from baseline).
Trough FEV1 | 4 weeks
  2. FEV1(L) measured in the morning prior to the dosing of inhaled medications on the last day of a 4-week (28 days) treatment (trough FEV1) after adjustment for baseline (change from baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Kostikas, Professor, Principal Investigator — University of Ioannina School of Medicine
Locations (1):
- BECRO Ltd., Athens, Greece